CLINICAL TRIAL: NCT03173976
Title: Anti-Osteoclast Therapy as Neoadjuvant in Treatment of Chondrosarcoma - Phase 1b Trial
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mohammed Milhem (Other)
Collaborators: Rising Tide Foundation (Other)
Responsible Party: Sponsor-Investigator, Mohammed Milhem, Clinical Professor Hematology/Oncology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201610743
Record Dates: First submitted 2017-05-29; First posted 2017-06-02 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Chondrosarcoma
MeSH Terms: conditions — Chondrosarcoma | interventions — Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: This is a single arm open label phase 1b clinical trial assessing the safety and efficacy of neoadjuvant zoledronic acid in patients with resectable any grade chondrosarcoma as measured by pathological characteristics and recurrence free survival.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zoledronic Acid (Experimental): 1 cycle of Zoledronic Acid (ZA) at 4mg IVP prior to surgery and a second cycle of ZA at 4 mg IVP 3 weeks after surgery
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid — Zoledronic acid, a member of bisphosphonate class, inhibits bone resorption.
  Other Names: Zometa®

SUMMARY:
The purpose of this single arm open label phase 1b clinical study is to see what effect zoledronic acid has on tumors in patients with resectable any grade chondrosarcoma prior to surgery.

DETAILED DESCRIPTION:
This is a single arm open label phase 1b clinical trial assessing the safety and efficacy of neoadjuvant zoledronic acid in patients with resectable any grade chondrosarcoma as measured by pathological characteristics and recurrence free survival. Prior to surgery, subjects will receive 1 standard dose of IV zoledronic acid given over 15 minutes. Surgery will be performed 21-31 days after the dose as per standard of care. The second standard dose of zoledronic acid will be given 3 weeks after surgery.

Phase 1b:

The Phase 1b portion of this study is to ensure the safety and tolerability of standard dose of zoledronic acid intravenously as assessed by incidence of dose limiting toxicities (DLT). Although the safety of use of this drug has been established in patients with bone metastases from solid tumors (breast, prostate) and in patients with hypercalcemia of malignancy and multiple myeloma, it has not been tested in patients with chondrosarcoma. Surgery will be performed between day 21 to 31 from the dose of zoledronic acid to allow its effect on the tumor and resolution of toxicities. A total of 6 patients will be enrolled in this run-in phase 1b. Patients will be followed post operatively as per NCCN guidelines (for years 1 and 2) with local and systemic imaging.

Expansion Cohort:

The phase 1 b expansion cohort of the study will provide an estimate of the relative treatment effect of zoledronic acid on any grade chondrosarcoma specimens. Subjects will receive a total of 2 doses of zoledronic acid, one dose prior to surgery and the second dose 21 days after surgery. Patients will undergo standard of care surgery 21-31 days from the first dose of zoledronic acid. 9 subjects will be enrolled in this cohort for a total of 15 planned subject enrollment over 3 years. Patients will be followed post operatively for recurrence with imaging and survival and as per NCCN guidelines (for years 1 and 2).

ELIGIBILITY:
Inclusion criteria

1. Male or female patients aged >/= 18 years old
2. ECOG Performance Status of </= 2
3. Written informed consent from subject or the subject's legally authorized representative, obtained prior to participation in the study and any related procedures being performed
4. Patients must meet the following laboratory criteria:

   1. Hematology:

      * Neutrophil count of >1500/mm
      * Platelet count of > 100,000/mm3
      * Hemoglobin ≥ 9 g/dL
   2. Biochemistry:

      * AST/SGOT and ALT/SGPT </=2.5 x upper limit of normal (ULN) or </=5.0 x ULN if the transaminase elevation is due to disease involvement
      * Serum bilirubin </= 1.5 x ULN; for subjects with Gilbert's syndrome, direct bilirubin </=1.5×ULN and indirect bilirubin </=3×ULN
      * Serum creatinine </= 1.5 x ULN or estimated creatinine clearance >/= 50 ml/min by Cockcroft-Gault equation: GFR=(140-age)*(wt in kg)*(0.85 if female)/(72xCr)
      * Total serum calcium (corrected for serum albumin) >/= 8.5 mg/dL or ionized calcium >/= 3.8 mg/dL
      * Serum potassium >/= LLN
      * Serum sodium >/= LLN
      * Serum albumin >/= 3g/dl
5. Any patient with a biopsy proven diagnosis of chondrosarcoma that is grade I, II or III or in cases where histological and radiological correlation suggests low grade chondrosarcoma as per multidisciplinary discussion.
6. Patients with biopsy proven dedifferentiated chondrosarcoma that chose not to pursue neoadjuvant chemotherapy are allowed.
7. Patients must not have received zoledronic acid (ZA) for any reason prior to the study.
8. Patients with metastatic disease are allowed, if indication to remove primary tumor.

Exclusion criteria

1. Prior use of Osteoclast inhibitors for osteoporosis within 6 months from screening will not be allowed.
2. Impaired cardiac function
3. Uncontrolled hypertension
4. Creatinine >1.5 or history of Renal disease preventing use of ZA.
5. Other concurrent severe and/or uncontrolled medical conditions including need for urgent dentoalveolar surgery as indicated by preventative dental exam
6. Concomitant use of any anti-cancer therapy or radiation therapy
7. Women who are pregnant or breast feeding or WOCBP not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1b cohort: Dose Limiting Toxicity - to examine the toxicity related to the therapy by measuring the number of treatment related adverse events in patients | All eligible patients that have initiated treatment will be considered evaluable for assessing adverse event rate(s) up to 4 weeks post Cycle 2
  Toxicity will be assessed using the NIH-NCI Common Terminology Criteria for Adverse Events, version 4.0 (CTCAEv4.)
Expansion cohort: Response Rate - Change at evaluations | Changes on 2 consecutive evaluations at screening phase (days 1-14); Cycle 2 at 3 weeks post operatively; EOT visit at 4 weeks post Cycle 2; and then at follow up visits every 6 months for up to 5 years.
  Response and progression will be assessed by tumor viability, osteoclast activity, and bone destruction compared to the initial biopsy in subjects with localized any grade chondrosarcoma.

SECONDARY OUTCOMES:
Recurrence (local or metastatic) free survival | All eligible patients that have initiated treatment will be considered evaluable for assessing recurrence free survival for up to 2 years.
  Recurrence-free survival will be estimated using the Kaplan-Meier method.
Overall survival | All eligible patients that have initiated treatment will be considered evaluable for assessing overall survival up to 5 years.
  Overall survival will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milhem, MBBS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No